CLINICAL TRIAL: NCT03580967
Title: Vortioxetine Monotherapy for Major Depressive Disorder in Type 2 Diabetes: Role of Inflammation, Kynurenine Pathway, and Structural and Functional Brain Connectivity as Biomarkers
Brief Title: Vortioxetine Monotherapy for Major Depressive Disorder in Type 2 Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 Pandemic interfered with Pt recruitment
Sponsor: Todd Doyle (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Todd Doyle, Assistant Professor, Loyola University
Organization: Loyola University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210161
Record Dates: First submitted 2018-06-25; First posted 2018-07-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Type2 Diabetes; Major Depressive Disorder
Keywords: Type 2 Diabetes; Major Depressive Disorder; Vortioxetine
MeSH Terms: conditions — Depressive Disorder, Major; Diabetes Mellitus, Type 2 | interventions — Vortioxetine

STUDY DESIGN:
Intervention Model Description: All participants will receive a 10 or 20 mg dose of vortioxetine to take daily for 8 weeks. Study PI and sub-investigator (psychiatrist Murali Rao, MD) will determine appropriate dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug: Vortioxetine (Other)
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Oral pill to be taken daily for 8 weeks, 10 or 20 mg dosage. Participants who cannot tolerate this dose may be reduced to 5mg dose.
  Other Names: Trintellix

SUMMARY:
This study will enroll participants who have been diagnosed with type 2 diabetes and are experiencing symptoms of depression. This study will look at an anti-depressant medication called vortioxetine (Trintellix). Vortioxetine is an oral medication (pill) that has been approved by the US Food and Drug Administration (FDA) to treat depression in adults.

The purpose of this study is to look at what effects (if any) vortioxetine may have on symptoms of depression in patients with type 2 diabetes. This study will also look at what effects (if any) vortioxetine has on blood sugar, and how vortioxetine may improve the way our brains are able to adapt and respond to stress.

DETAILED DESCRIPTION:
This will be a 9-week, open-label, single-arm, pilot investigation for Type 2 Diabetes (T2D) patients with Major Depressive Disorder (MDD). The study includes a screening visit, a 1-week washout phase (or 30-day washout phase for serotonergic agents), and an 8-week flexible dose phase that includes the baseline and post-treatment follow-up visits. A minimum of N=70 participants will be enrolled in the treatment.

At the screening visit, the study will be explained and the informed consent process will take place. Patients who sign the IRB-approved consent form will undergo a psychiatric interview. The diagnosis of MDD will be established in this examination using the psychiatric interview and Hamilton Depression Rating Scale (HAM-D) by the study PI.

Eligible participants will be instructed how to taper the antidepressant they have been taking (if relevant) over the course of the one-week (or 30-days for serotonergic agents).

After these tapers, all participants will return for a baseline visit where they will be re-assessed to ensure persistent depressive symptoms. If patients continue to score ≥18 on the HAM-D, they will complete the psychosocial questionnaires; patients scoring below <18 on the HAM-D at this visit will be terminated from the study and offered conventional, standard of care treatment within LUMC Department of Psychiatry. Once participants are given the psychosocial questionnaires as part of the baseline visit, a blood draw will be conducted by the Study Nurse/Coordinator, and MRI scans will be completed.

At the end of the baseline session, participants will receive Vortioxetine for the remaining 8-week flexible dosing period (i.e., 10 mg to 20 mg dosing). In the instance a patient is unable to tolerate either 10 mg to 20 mg of Vortioextine (as reported in the medication packet insert), the patient will be allowed to reduce their dosage to 5 mg, which will be done in consultation with the PI and sub-investigator.

Following the 8-week intervention, participants will be scheduled for the post visit, which will include the following: another clinical interview and HAM-D conducted by the PI, completion of post visit-related psychosocial questionnaires, a second blood draw conducted by the Study Nurse/Coordinator, and then post visit-MRI scans will be completed. Should any patients continue to score >18 on the HAM-D at study conclusion, resources and referrals will be provided for further psychological/psychiatric interventions, as needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40 to 65 years of age at time of screening visit.
* Women only: Must be post-menopausal at time of screening visit (i.e., defined by NO menstruation for at least the past 12-months).
* Diagnosis of T2D, as defined by a diagnosis of T2D (for at least 12 months) in the medical record made by a physician (i.e., denoted as 250.XX according to ICD-9/ICD-10 billing codes) OR
* current use of oral hypoglycemic medications or insulin OR
* having a fasting plasma glucose ≥126 mg/dL in the medical record OR
* having a 2-hour oral glucose tolerance test ≥200 mg/dL in the medical record
* Patients who meet criteria for current MDD without significant co-morbid psychiatric diagnoses, as determined by study PI from screening visit:
* Clinical Psychiatric Interview to determine DSM-V criteria for current MDD AND
* A minimum score of 18 on the Hamilton Depression Scale (HAM-D)
* Patients with T2D and current MDD that would benefit from antidepressant therapy, which may include:
* Patients with current MDD who were NOT prescribed an antidepressant medication in the past;
* Patients with current MDD who are NOT responding to their current prescribed antidepressant;
* Patients with current MDD who are experiencing breakthrough depressive symptoms despite being maintained on another antidepressant.
* Must have the ability to provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with any form of contraindication to Vortioxetine treatment, as outlined in the medication packet insert, (e.g., presence of a known hypersensitivity to the study drug or hypersensitivity to MAO-I use, etc.).

MRI-Related Exclusion Criteria

* Participants weighing >550 lbs (per MRI weight restrictions set by Loyola University Medical Center);
* Patients with a pacemaker, AICD, ossicular prosthesis, nerve stimulator, or another contraindication to MRI;
* Pregnant patients;
* Patients with an inability to tolerate being in enclosed places/spaces such as MRI;
* Patients with a history of neurosurgery, brain irradiation, or cerebral endovascular treatment.;
* Patients with history of epilepsy, stroke, neurodegenerative disorder, severe traumatic brain injury, hydrocephalus or demyelinating disorder;
* Patients with a history of malignant neoplasm

Exclusion Criteria to Reduce False Positive Rates of Inflammation

* Specific pre-existing chronic pain conditions such as rheumatoid arthritis or fibromyalgia. However, this will NOT include more localized pain-related conditions such as low-back pain or complications associated with T2D (e.g., diabetic neuropathy).
* History of peptic ulcer complicated by perforation, hemorrhage, or obstruction; symptoms of peptic ulcer within 4 weeks of enrollment date that has not been treated.
* Current diagnosis of substance abuse/dependence during the 6 months prior to study enrollment.
* Current diagnosis of uncontrolled hypertension, anemia, liver disease, kidney disease, stroke, and autoimmune disease. Based on the clinical judgment of the study PI, a risk assessment will be conducted if a participant endorses any of these diagnoses but would be otherwise a suitable participant to enroll in the study.
* Current acute infection/infectious disease (i.e., a cold or the flu). Based on the clinical judgement of the study PI, a risk assessment will be conducted if a participant endorses some acute infection/infectious disease, but would be otherwise suitable to enroll in the study following a brief wait period for full symptom remission.
* Pre- and peri-menopausal women (i.e., defined as the presence of ANY menstruation within the past 12 months).
* Certain steroids (e.g., use of hormonal birth control) and any systemic corticosteroids. Please note that hormone replacement therapy will be allowed along with any topical corticosteroid creams.
* Patients currently enrolled in any other clinical trial for treatment of MDD (e.g., patients receiving experimental vitamin D supplementation).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms measured by Hamilton Depression Rating Scale (HAM-D) | Baseline and End of Treatment visit (Week 8)
  The HAM-D is an 18-item questionnaire used to provide an indication of depression. The patient is rated by a clinician on 18 items scored on a 3-point or 5-point Likert-type scale. Remission of Major Depressive Disorder symptoms is defined as a total score on the HAM-D of ≤ 7.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Doyle, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention, National Diabetes Statistics Report. National diabetes statistics report. https://www.cdc.gov/diabetes/pdfs/data/statistics/national-diabetes-statistics-report.pdf. (2017).
- [Background] Anderson RJ, Freedland KE, Clouse RE, Lustman PJ. The prevalence of comorbid depression in adults with diabetes: a meta-analysis. Diabetes Care. 2001 Jun;24(6):1069-78. doi: 10.2337/diacare.24.6.1069. PMID 11375373
- [Background] Gavard JA, Lustman PJ, Clouse RE. Prevalence of depression in adults with diabetes. An epidemiological evaluation. Diabetes Care. 1993 Aug;16(8):1167-78. doi: 10.2337/diacare.16.8.1167. PMID 8375247
- [Background] de Groot M, Doyle T, Hockman E, Wheeler C, Pinkerman B, Shubrook J, Gotfried R, Schwartz F. Depression among type 2 diabetes rural Appalachian clinic attendees. Diabetes Care. 2007 Jun;30(6):1602-4. doi: 10.2337/dc06-1599. Epub 2007 Mar 12. No abstract available. PMID 17353505
- [Background] Lustman PJ, Anderson RJ, Freedland KE, de Groot M, Carney RM, Clouse RE. Depression and poor glycemic control: a meta-analytic review of the literature. Diabetes Care. 2000 Jul;23(7):934-42. doi: 10.2337/diacare.23.7.934. PMID 10895843
- [Background] de Groot M, Anderson R, Freedland KE, Clouse RE, Lustman PJ. Association of depression and diabetes complications: a meta-analysis. Psychosom Med. 2001 Jul-Aug;63(4):619-30. doi: 10.1097/00006842-200107000-00015. PMID 11485116
- [Background] Ciechanowski PS, Katon WJ, Russo JE. Depression and diabetes: impact of depressive symptoms on adherence, function, and costs. Arch Intern Med. 2000 Nov 27;160(21):3278-85. doi: 10.1001/archinte.160.21.3278. PMID 11088090
- [Background] Jacobson AM, de Groot M, Samson JA. The effects of psychiatric disorders and symptoms on quality of life in patients with type I and type II diabetes mellitus. Qual Life Res. 1997 Jan;6(1):11-20. doi: 10.1023/a:1026487509852. PMID 9062437
- [Background] Egede LE, Osborn CY. Role of motivation in the relationship between depression, self-care, and glycemic control in adults with type 2 diabetes. Diabetes Educ. 2010 Mar-Apr;36(2):276-83. doi: 10.1177/0145721710361389. Epub 2010 Feb 23. PMID 20179250
- [Background] Katon W, von Korff M, Ciechanowski P, Russo J, Lin E, Simon G, Ludman E, Walker E, Bush T, Young B. Behavioral and clinical factors associated with depression among individuals with diabetes. Diabetes Care. 2004 Apr;27(4):914-20. doi: 10.2337/diacare.27.4.914. PMID 15047648
- [Background] Katon WJ, Rutter C, Simon G, Lin EH, Ludman E, Ciechanowski P, Kinder L, Young B, Von Korff M. The association of comorbid depression with mortality in patients with type 2 diabetes. Diabetes Care. 2005 Nov;28(11):2668-72. doi: 10.2337/diacare.28.11.2668. PMID 16249537
- [Background] Egede LE, Zheng D, Simpson K. Comorbid depression is associated with increased health care use and expenditures in individuals with diabetes. Diabetes Care. 2002 Mar;25(3):464-70. doi: 10.2337/diacare.25.3.464. PMID 11874931
- [Background] Baumeister H, Hutter N, Bengel J. Psychological and pharmacological interventions for depression in patients with diabetes mellitus and depression. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD008381. doi: 10.1002/14651858.CD008381.pub2. PMID 23235661
- [Background] van der Feltz-Cornelis CM, Nuyen J, Stoop C, Chan J, Jacobson AM, Katon W, Snoek F, Sartorius N. Effect of interventions for major depressive disorder and significant depressive symptoms in patients with diabetes mellitus: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):380-95. doi: 10.1016/j.genhosppsych.2010.03.011. Epub 2010 May 15. PMID 20633742
- [Background] Champaneri S, Wand GS, Malhotra SS, Casagrande SS, Golden SH. Biological basis of depression in adults with diabetes. Curr Diab Rep. 2010 Dec;10(6):396-405. doi: 10.1007/s11892-010-0148-9. PMID 20878274
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Stuart MJ, Baune BT. Depression and type 2 diabetes: inflammatory mechanisms of a psychoneuroendocrine co-morbidity. Neurosci Biobehav Rev. 2012 Jan;36(1):658-76. doi: 10.1016/j.neubiorev.2011.10.001. Epub 2011 Oct 14. PMID 22020230
- [Background] Pickup JC. Inflammation and activated innate immunity in the pathogenesis of type 2 diabetes. Diabetes Care. 2004 Mar;27(3):813-23. doi: 10.2337/diacare.27.3.813. PMID 14988310
- [Background] de Jonge P, Rosmalen JG. Comment on: Knol MJ, Twisk JWR, Beekman ATF, Heine RJ, Snoek FJ, Pouwer F. (2006) depression as a risk factor for the onset of type 2 diabetes mellitus. A meta-analysis. Diabetologia; 49: 837-845. Diabetologia. 2006 Nov;49(11):2797-8; author reply 2799-800. doi: 10.1007/s00125-006-0389-y. Epub 2006 Aug 18. No abstract available. PMID 16917758
- [Background] Ruhe HG, Mason NS, Schene AH. Mood is indirectly related to serotonin, norepinephrine and dopamine levels in humans: a meta-analysis of monoamine depletion studies. Mol Psychiatry. 2007 Apr;12(4):331-59. doi: 10.1038/sj.mp.4001949. Epub 2007 Jan 16. PMID 17389902
- [Background] Raison CL, Capuron L, Miller AH. Cytokines sing the blues: inflammation and the pathogenesis of depression. Trends Immunol. 2006 Jan;27(1):24-31. doi: 10.1016/j.it.2005.11.006. Epub 2005 Nov 28. PMID 16316783
- [Background] Doyle TA, de Groot M, Harris T, Schwartz F, Strotmeyer ES, Johnson KC, Kanaya A. Diabetes, depressive symptoms, and inflammation in older adults: results from the Health, Aging, and Body Composition Study. J Psychosom Res. 2013 Nov;75(5):419-24. doi: 10.1016/j.jpsychores.2013.08.006. Epub 2013 Aug 16. PMID 24182629
- [Background] Alvarez A, Faccioli J, Guinzbourg M, Castex MM, Bayon C, Masson W, Bluro I, Kozak A, Sorroche P, Capurro L, Grosembacher L, Proietti A, Finkelsztein C, Costa L, Fainstein Day P, Cagide A, Litwak LE, Golden SH. Endocrine and inflammatory profiles in type 2 diabetic patients with and without major depressive disorder. BMC Res Notes. 2013 Feb 14;6:61. doi: 10.1186/1756-0500-6-61. PMID 23410093
- [Background] Hood KK, Lawrence JM, Anderson A, Bell R, Dabelea D, Daniels S, Rodriguez B, Dolan LM; SEARCH for Diabetes in Youth Study Group. Metabolic and inflammatory links to depression in youth with diabetes. Diabetes Care. 2012 Dec;35(12):2443-6. doi: 10.2337/dc11-2329. Epub 2012 Oct 1. PMID 23033243
- [Background] Yoshimura R, Hori H, Ikenouchi-Sugita A, Umene-Nakano W, Ueda N, Nakamura J. Higher plasma interleukin-6 (IL-6) level is associated with SSRI- or SNRI-refractory depression. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Jun 15;33(4):722-6. doi: 10.1016/j.pnpbp.2009.03.020. Epub 2009 Mar 28. PMID 19332097
- [Background] Myint AM, Kim YK. Cytokine-serotonin interaction through IDO: a neurodegeneration hypothesis of depression. Med Hypotheses. 2003 Nov-Dec;61(5-6):519-25. doi: 10.1016/s0306-9877(03)00207-x. PMID 14592780
- [Background] Munipally PK, Agraharm SG, Valavala VK, Gundae S, Turlapati NR. Evaluation of indoleamine 2,3-dioxygenase expression and kynurenine pathway metabolites levels in serum samples of diabetic retinopathy patients. Arch Physiol Biochem. 2011 Dec;117(5):254-8. doi: 10.3109/13813455.2011.623705. Epub 2011 Oct 29. PMID 22034910
- [Background] Doyle T, Halaris A, Rao M. Shared neurobiological pathways between type 2 diabetes and depressive symptoms: a review of morphological and neurocognitive findings. Curr Diab Rep. 2014 Dec;14(12):560. doi: 10.1007/s11892-014-0560-7. PMID 25381209
- [Background] Fossati P, Radtchenko A, Boyer P. Neuroplasticity: from MRI to depressive symptoms. Eur Neuropsychopharmacol. 2004 Dec;14 Suppl 5:S503-10. doi: 10.1016/j.euroneuro.2004.09.001. PMID 15550349
- [Background] Reagan LP. Diabetes as a chronic metabolic stressor: causes, consequences and clinical complications. Exp Neurol. 2012 Jan;233(1):68-78. doi: 10.1016/j.expneurol.2011.02.004. Epub 2011 Feb 12. PMID 21320489
- [Background] Ho N, Sommers MS, Lucki I. Effects of diabetes on hippocampal neurogenesis: links to cognition and depression. Neurosci Biobehav Rev. 2013 Sep;37(8):1346-62. doi: 10.1016/j.neubiorev.2013.03.010. Epub 2013 May 13. PMID 23680701
- [Background] Maes M, Yirmyia R, Noraberg J, Brene S, Hibbeln J, Perini G, Kubera M, Bob P, Lerer B, Maj M. The inflammatory & neurodegenerative (I&ND) hypothesis of depression: leads for future research and new drug developments in depression. Metab Brain Dis. 2009 Mar;24(1):27-53. doi: 10.1007/s11011-008-9118-1. Epub 2008 Dec 16. PMID 19085093
- [Background] Koehl M, Abrous DN. A new chapter in the field of memory: adult hippocampal neurogenesis. Eur J Neurosci. 2011 Mar;33(6):1101-14. doi: 10.1111/j.1460-9568.2011.07609.x. PMID 21395854
- [Background] Snyder JS, Hong NS, McDonald RJ, Wojtowicz JM. A role for adult neurogenesis in spatial long-term memory. Neuroscience. 2005;130(4):843-52. doi: 10.1016/j.neuroscience.2004.10.009. PMID 15652983
- [Background] Ajilore O, Narr K, Rosenthal J, Pham D, Hamilton L, Watari K, Elderkin-Thompson V, Darwin C, Toga A, Kumar A. Regional cortical gray matter thickness differences associated with type 2 diabetes and major depression. Psychiatry Res. 2010 Nov 30;184(2):63-70. doi: 10.1016/j.pscychresns.2010.07.003. Epub 2010 Sep 15. PMID 20832254
- [Background] Kumar A, Gupta R, Thomas A, Ajilore O, Hellemann G. Focal subcortical biophysical abnormalities in patients diagnosed with type 2 diabetes and depression. Arch Gen Psychiatry. 2009 Mar;66(3):324-30. doi: 10.1001/archgenpsychiatry.2008.548. PMID 19255382
- [Background] Kumar A, Haroon E, Darwin C, Pham D, Ajilore O, Rodriguez G, Mintz J. Gray matter prefrontal changes in type 2 diabetes detected using MRI. J Magn Reson Imaging. 2008 Jan;27(1):14-9. doi: 10.1002/jmri.21224. PMID 18050330
- [Background] Awad N, Gagnon M, Messier C. The relationship between impaired glucose tolerance, type 2 diabetes, and cognitive function. J Clin Exp Neuropsychol. 2004 Nov;26(8):1044-80. doi: 10.1080/13803390490514875. PMID 15590460
- [Background] Connolly KR, Thase ME. Vortioxetine: a New Treatment for Major Depressive Disorder. Expert Opin Pharmacother. 2016;17(3):421-31. doi: 10.1517/14656566.2016.1133588. PMID 26679430
- [Background] Bang-Andersen B, Ruhland T, Jorgensen M, Smith G, Frederiksen K, Jensen KG, Zhong H, Nielsen SM, Hogg S, Mork A, Stensbol TB. Discovery of 1-[2-(2,4-dimethylphenylsulfanyl)phenyl]piperazine (Lu AA21004): a novel multimodal compound for the treatment of major depressive disorder. J Med Chem. 2011 May 12;54(9):3206-21. doi: 10.1021/jm101459g. Epub 2011 Apr 12. PMID 21486038
- [Background] Mork A, Pehrson A, Brennum LT, Nielsen SM, Zhong H, Lassen AB, Miller S, Westrich L, Boyle NJ, Sanchez C, Fischer CW, Liebenberg N, Wegener G, Bundgaard C, Hogg S, Bang-Andersen B, Stensbol TB. Pharmacological effects of Lu AA21004: a novel multimodal compound for the treatment of major depressive disorder. J Pharmacol Exp Ther. 2012 Mar;340(3):666-75. doi: 10.1124/jpet.111.189068. Epub 2011 Dec 9. PMID 22171087
- [Background] Westrih I, Rehrson A, & Zhong H, et al. In vitro and in vivo effects for the multimodal antidepressant vortioxetine (Lu AA21004) at human and rat targets. International Journal of Psychiatry and Clinical Practice 2012; 16 (S1): 47.
- [Background] Florea I, Loft H, Danchenko N, Rive B, Brignone M, Merikle E, Jacobsen PL, Sheehan DV. The effect of vortioxetine on overall patient functioning in patients with major depressive disorder. Brain Behav. 2017 Feb 2;7(3):e00622. doi: 10.1002/brb3.622. eCollection 2017 Mar. PMID 28293465
- [Background] McIntyre RS, Harrison J, Loft H, Jacobson W, Olsen CK. The Effects of Vortioxetine on Cognitive Function in Patients with Major Depressive Disorder: A Meta-Analysis of Three Randomized Controlled Trials. Int J Neuropsychopharmacol. 2016 Jun 15;19(10):pyw055. doi: 10.1093/ijnp/pyw055. PMID 27312740
- [Background] Nomikos GG, Tomori D, Zhong W, Affinito J, Palo W. Efficacy, safety, and tolerability of vortioxetine for the treatment of major depressive disorder in patients aged 55 years or older. CNS Spectr. 2017 Aug;22(4):348-362. doi: 10.1017/S1092852916000626. Epub 2016 Nov 21. PMID 27869048
- [Background] de Groot M, Doyle T, Kushnick M, Shubrook J, Merrill J, Rabideau E, Schwartz F. Can lifestyle interventions do more than reduce diabetes risk? Treating depression in adults with type 2 diabetes with exercise and cognitive behavioral therapy. Curr Diab Rep. 2012 Apr;12(2):157-66. doi: 10.1007/s11892-012-0261-z. PMID 22350739
- [Background] Calabrese JR, Skwerer RG, Barna B, Gulledge AD, Valenzuela R, Butkus A, Subichin S, Krupp NE. Depression, immunocompetence, and prostaglandins of the E series. Psychiatry Res. 1986 Jan;17(1):41-7. doi: 10.1016/0165-1781(86)90040-5. PMID 2935897
- [Background] Funakoshi-Tago M, Shimizu T, Tago K, Nakamura M, Itoh H, Sonoda Y, Kasahara T. Celecoxib potently inhibits TNFalpha-induced nuclear translocation and activation of NF-kappaB. Biochem Pharmacol. 2008 Sep 1;76(5):662-71. doi: 10.1016/j.bcp.2008.06.015. Epub 2008 Jul 3. PMID 18644347
- [Background] Hayashino Y, Mashitani T, Tsujii S, Ishii H; Diabetes Distress and Care Registry at Tenri Study Group. Elevated levels of hs-CRP are associated with high prevalence of depression in japanese patients with type 2 diabetes: the Diabetes Distress and Care Registry at Tenri (DDCRT 6). Diabetes Care. 2014 Sep;37(9):2459-65. doi: 10.2337/dc13-2312. Epub 2014 Jun 26. PMID 24969579
- [Background] Husain MM, Rush AJ, Trivedi MH, McClintock SM, Wisniewski SR, Davis L, Luther JF, Zisook S, Fava M. Pain in depression: STAR*D study findings. J Psychosom Res. 2007 Aug;63(2):113-22. doi: 10.1016/j.jpsychores.2007.02.009. PMID 17662746
- [Background] Lanquillon S, Krieg JC, Bening-Abu-Shach U, Vedder H. Cytokine production and treatment response in major depressive disorder. Neuropsychopharmacology. 2000 Apr;22(4):370-9. doi: 10.1016/S0893-133X(99)00134-7. PMID 10700656
- [Background] Leuchter AF, Husain MM, Cook IA, Trivedi MH, Wisniewski SR, Gilmer WS, Luther JF, Fava M, Rush AJ. Painful physical symptoms and treatment outcome in major depressive disorder: a STAR*D (Sequenced Treatment Alternatives to Relieve Depression) report. Psychol Med. 2010 Feb;40(2):239-51. doi: 10.1017/S0033291709006035. Epub 2009 Jun 3. PMID 19493369
- [Background] Lieb J, Karmali R, Horrobin D. Elevated levels of prostaglandin E2 and thromboxane B2 in depression. Prostaglandins Leukot Med. 1983 Apr;10(4):361-7. doi: 10.1016/0262-1746(83)90048-3. PMID 6574523
- [Background] Miller CL, Llenos IC, Dulay JR, Weis S. Upregulation of the initiating step of the kynurenine pathway in postmortem anterior cingulate cortex from individuals with schizophrenia and bipolar disorder. Brain Res. 2006 Feb 16;1073-1074:25-37. doi: 10.1016/j.brainres.2005.12.056. Epub 2006 Jan 30. PMID 16448631
- [Background] Miller GE, Rohleder N, Cole SW. Chronic interpersonal stress predicts activation of pro- and anti-inflammatory signaling pathways 6 months later. Psychosom Med. 2009 Jan;71(1):57-62. doi: 10.1097/PSY.0b013e318190d7de. Epub 2008 Dec 10. PMID 19073750
- [Background] Myint AM, Kim YK, Verkerk R, Park SH, Scharpe S, Steinbusch HW, Leonard BE. Tryptophan breakdown pathway in bipolar mania. J Affect Disord. 2007 Sep;102(1-3):65-72. doi: 10.1016/j.jad.2006.12.008. Epub 2007 Jan 30. PMID 17270276
- [Background] Myint AM, Kim YK, Verkerk R, Scharpe S, Steinbusch H, Leonard B. Kynurenine pathway in major depression: evidence of impaired neuroprotection. J Affect Disord. 2007 Feb;98(1-2):143-51. doi: 10.1016/j.jad.2006.07.013. Epub 2006 Sep 6. PMID 16952400
- [Background] O'Brien SM, Scully P, Fitzgerald P, Scott LV, Dinan TG. Plasma cytokine profiles in depressed patients who fail to respond to selective serotonin reuptake inhibitor therapy. J Psychiatr Res. 2007 Apr-Jun;41(3-4):326-31. doi: 10.1016/j.jpsychires.2006.05.013. Epub 2006 Jul 25. PMID 16870211
- [Background] Pilowsky I, Spence N, Cobb J, Katsikitis M. The Illness Behavior Questionnaire as an aid to clinical assessment. Gen Hosp Psychiatry. 1984 Apr;6(2):123-30. doi: 10.1016/0163-8343(84)90070-7. PMID 6714666
- [Background] Riondino S, Trifiro E, Principessa L, Mascioletti S, Di Renzo L, Gaudio C, Biasucci LM, Crea F, Pulcinelli FM. Lack of biological relevance of platelet cyclooxygenase-2 dependent thromboxane A2 production. Thromb Res. 2008;122(3):359-65. doi: 10.1016/j.thromres.2007.12.011. Epub 2008 Mar 4. PMID 18295304
- [Background] Rosenbaum D, Haipt A, Fuhr K, Haeussinger FB, Metzger FG, Nuerk HC, Fallgatter AJ, Batra A, Ehlis AC. Aberrant functional connectivity in depression as an index of state and trait rumination. Sci Rep. 2017 May 19;7(1):2174. doi: 10.1038/s41598-017-02277-z. PMID 28526867
- [Background] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Background] Cohen, J. (1988). Statistical Power Analyses for the Behavioral Sciences (2nd Edition). Psychology Press. Taylor & Francis Group.
- [Background] de Groot M, Doyle T, Averyt J, Risaliti C, Shubroo J. Depressive symptoms and type 2 diabetes mellitus in rural appalachia: an 18-month follow-up study. Int J Psychiatry Med. 2015;48(4):263-77. doi: 10.2190/PM.48.4.c. PMID 25817523